CLINICAL TRIAL: NCT00150163
Title: Odense Androgen Study - A Population-Based Study of Androgens, Body Composition, and Muscle Function in 20-29 Year-Old Danish Men
Brief Title: Odense Androgen Study: Study of Androgens, Body Composition, and Muscle Function in Danish Men
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Other Study IDs: 015
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2005-09

CONDITIONS: Bone Diseases
Keywords: Androgens; Bone; Muscle; Estrogens; Fat; Lipid and glucose metabolism
MeSH Terms: conditions — Bone Diseases; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objective:

* To define a reference-population of healthy young men (20-29 years old).
* To establish reference-intervals for:

  1. Total, bioavailable and free serum androgens (testosterone, dihydrotestosterone, androstenedione) and serum estrogens (estradiol, estrone).
  2. Total and free IGF-1.
* To study the influence of physical activity, alcohol intake, tobacco and abuse of anabolic steroids on serum levels of androgens.
* To identify the androgens (or estrogens) that primarily reflect the following parameters:

  1. Muscle mass, muscle strength, muscle power, oxygen uptake, and hematocrit.
  2. Bone mineral density and bone metabolism.
  3. Total and visceral fat mass.
  4. Lipid- and glucose metabolism and glucocorticoid metabolism.
  5. Sexual function and quality of life.
* To study the modifying effect of birth weight, the AR gene CAG-repeat polymorphism, and the level of IGF-1 on associations between serum androgens and the measures above:

Ethics, design and schedule:

The local ethic review board approved a population-based, cross-sectional study planned for the inclusion of 800 Caucasian men, 20 to 29 year old, living in the County of Funen. The only exclusion criteria were opioid drug addiction, cancer, and severe chronic disease. A basic questionnaire was mailed to 3000 men, randomly drawn from the Danish Central Personal Registry. Adequately answered questionnaires were returned from 2,199 men, who subsequently received an invitation to participate. Informed consent was obtained from 783 men. The examinations started in March 2002 and terminated in May 2003. Within subject variation was determined for all study parameters in 20 men. The men included matched the men answering the questionnaire on all questionnaire items and demographics. All analyses have been performed, except for the additional serum sex hormone assays, IGF-1 assays and AR gene analyses.

A sequential rule-out from the reference population was performed on the following criteria:

1. testicular pathology: bilateral cryptorchidism, varicocele, testes volumina < 10 ml (each), history of spermatic cord torsion.
2. severe chronic disease.
3. regular medication or abuse of anabolic steroids.
4. body mass index < 19 kg/m2.
5. safety serum parameters: luteinizing hormone (LH) <1.0 U/L or >8.4 U/l, alanine-amino-transferase (ALAT) >70 U/l and thyrotropin (TSH) >6.0 mU/l.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-29 years
* Residence: County of Funen, Denmark

Exclusion Criteria:

* Opioid drug addiction
* Cancer
* Severe chronic disease

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800
Dates: Start 2002-03; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Torben L. Nielsen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Result] Nielsen TL, Wraae K, Brixen K, Hermann AP, Andersen M, Hagen C. Prevalence of overweight, obesity and physical inactivity in 20- to 29-year-old, Danish men. Relation to sociodemography, physical dysfunction and low socioeconomic status: the Odense Androgen Study. Int J Obes (Lond). 2006 May;30(5):805-15. doi: 10.1038/sj.ijo.0803197. PMID 16418764
- [Derived] Frost M, Abrahamsen B, Nielsen TL, Hagen C, Andersen M, Brixen K. Vitamin D status and PTH in young men: a cross-sectional study on associations with bone mineral density, body composition and glucose metabolism. Clin Endocrinol (Oxf). 2010 Nov;73(5):573-80. doi: 10.1111/j.1365-2265.2010.03847.x. PMID 20718769